CLINICAL TRIAL: NCT03333187
Title: Ruxolitinib Versus Allogeneic Stem Cell Transplantation for Patients With Myelofibrosis According to Donor Availability: A Prospective Phase II Trial (MMM 02 Study)
Brief Title: Ruxolitinib vs Allogeneic SCT for Patients With Myelofibrosis According to Donor Availability
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Novartis (Industry); Clinical Trial Center North (CTC North GmbH & Co. KG) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMM 02 study / RuxoAlloStudy
Record Dates: First submitted 2017-06-22; First posted 2017-11-06 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Bone Marrow Fibrosis
Keywords: Myelofibrosis, Myeloproliferative Disease
MeSH Terms: conditions — Primary Myelofibrosis; Myeloproliferative Disorders | interventions — ruxolitinib

STUDY DESIGN:
Intervention Model Description: Treatment A (only with a suitable stem cell donor):
  Allogeneic SCT after 3 months of Ruxolitinib induction therapy
  Treatment B:
  Ruxolitinib continuous therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Treatment with Allogeneic Stem cell Transplantation after 3 months of Ruxolitinib induction therapy
  Interventions: Procedure: Allogeneic stem cell transplantation
- Arm B (Active Comparator): Treatment with Ruxolitinib continuous therapy
  Interventions: Drug: Ruxolitinib continuous therapy

INTERVENTIONS:
Procedure: Allogeneic stem cell transplantation
  Arms: Arm A
Drug: Ruxolitinib continuous therapy
  Other Names: Jakavi
  Arms: Arm B

SUMMARY:
The present study will be a multicenter, prospective phase II-study comparing efficacy of allogeneic SCT for patients with myelofibrosis who have a suitable stem cell donor after a 3 months Ruxolitinib induction therapy with patients who lack a suitable stem cell donor and will continue to receive Ruxolitinib.

DETAILED DESCRIPTION:
This study is a multicenter, prospective phase II-study compares efficacy of allogeneic SCT for patients with myelofibrosis who have a suitable stem cell donor after a 3 months Ruxolitinib induction therapy with patients who lack a suitable stem cell donor and will continue to receive Ruxolitinib.

In this study will further assess and compare the safety and efficacy of study treatments/ induction therapy in both study arms on spleen reduction, improvement of constitutional symptoms, QOL, toxicity, fibrosis regression, development of GvHD as well as chimerism, engraftment, relapse incidence, disease related mortality, outcome and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic primary myelofibrosis or myelofibrosis post polycythaemia vera or essential thrombocythemia stage intermediate 2- or high-risk according to IPSS or DIPSS [46] or intermediate 1-risk with high risk cytogenetics, other than normal karyotype, sole del 20q, del 13q, or sole+9, or transfusion-dependency
2. Patients age: 18 - 70 years at time of inclusion (female and male)
3. Patients understand and voluntarily sign an informed consent form
4. Platelet count ≥ 50 x 109/L
5. No prior Ruxolitinib treatment
6. ECOG ≤ 2

Exclusion Criteria:

1. Severe renal, hepatic, pulmonary or cardiac disease, such as:

   * Total bilirubin, SGPT or SGOT > 3 times upper the normal level
   * Left ventricular ejection fraction < 30 %
   * Creatinine clearance < 30 ml/min
   * DLCO < 35 % and/or receiving supplementary continuous oxygen
2. Positive serology for HIV
3. Pregnant or lactating women (positive serum pregnancy test)
4. Age < 18 and ≥ 71 years.
5. Uncontrolled invasive fungal infection at time of screening (baseline)
6. Serious psychiatric or psychological disorders
7. Participation in another study with ongoing use of unlicensed investigational product from 28 days before study enrollment
8. Transformation to AML

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2025-10-07 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 3 years
  Compare to event free survival of patients at 3 years after allogeneic SCT and in Ruxolitinib continuous therapy in patients without a suitable donor

SECONDARY OUTCOMES:
Spleen reduction | 3 months
  Ultrasound measurement Spleen size, reduction of Spleen size after 3 months Ruxolitinib induction therapy
Improvement of constitutional symptoms | 3 months
  Improvement of constitutional symptoms (Loose of weight and night sweat) after 3 months Ruxolitinib induction therapy, questionnaire, medical history
Improvement of bone marrow fibrosis | 3 months
  bone marrow histology, Improvement of bone marrow fibrosis after 3 months of Ruxolitinib induction therapy
Acute graft-versus-host disease | Day +100 after allogeneic SCT
  Incidence of acute graft-versus-host disease on Day +100 after allogeneic SCT according to the Glucksberg scale revised by Przepiorka
Chronic graft-versus-host disease | 1, 2 and 3 years after allogeneic SCT
  Incidence of chronic graft-versus-host disease according to the NIH consensus criteria of Filipovich et al. at 1, 2 and 3 years after allogeneic SCT
Toxicity of Ruxolitinib | till 3 years
  Toxicity of Ruxolitinib scored according to NCI CTCAE, Version 4.0
Toxicity of conditioning therapy | till 3 years
  Toxicity of conditioning therapy scored according to NCI CTCAE, Version 4.0
Relapse | 3 years
  Cumulative incidence of relapse at 3 years after allogeneic SCT
Disease-related mortality | 3 years
  Disease-related mortality at 3 years after allogeneic SCT and Ruxolitinib continuous therapies
Non-relapsed mortality | 1 and 3 years
  Non-relapsed mortality at 1 and 3 years after allogeneic SCT and Ruxolitinib continuous therapy
Discontinuation rate | 3 years
  Discontinuation rate at 3 years after Ruxolitinib continuous therapy (End of study)
Evaluation of Sorror Risk Score | at baseline
  Evaluation of Sorror Risk Score on outcome after allogeneic SCT
Chimerism on relapse | 30d, 100d, 180 d, 1 year, 2 years and 3 years
  Chimerism Analyse, Impact of chimerism on relapse incidence after allogeneic SCT
Bone marrow fibrosis regression | 30d, 100d, 1 year, and 3 years
  bone marrow histology, Evaluation of bone marrow fibrosis regression after allogeneic SCT at 30d, 100d, 1 year, and 3 years
Bone marrow fibrosis regression | 30d, 100d, 1 year and 3 years
  bone marrow histology, Evaluation of bone marrow fibrosis regression after Ruxolitinib continuous therapy at 30d, 100d, 1 year and 3 years
Evaluation of QOL (FACT-BMT) | baseline, at transplantation, +180d, +1 year, +2 years and +3 years
  Questionnaire, Evaluation of QOL (FACT-BMT) before Ruxolitinib induction therapy (= baseline), at transplantation, and after transplantation at 6m, 1 year, 2 years and 3 years
Evaluation of QOL (MPN-SAF-TSS) | baseline, at transplantation, +180d, +1 year, +2 years and +3 years
  Questionaire, Evaluation of QOL (MPN-SAF-TSS) before Ruxolitinib induction therapy (= baseline), at transplantation, and after transplantation at 6m, 1 year, 2 years and 3 years
Evaluation of QOL (FACT-BMT) | baseline, confinement to Ruxolitinib continous therapy, +180d, +1 year, +2 years and +3 years
  Questionnaire, Evaluation of QOL (FACT-BMT) before Ruxolitinib induction therapy (= baseline), at confinement to Ruxolitinib continuous therapy and after confinement at 6 months, 1 year, 2 years and 3 years
Evaluation of QOL (MPN-SAF-TSS) | baseline, confinement to Ruxolitinib continous therapy, +180d, +1 year, +2 years and +3 years
  Questionnaire, Evaluation of QOL (MPN-SAF-TSS) before Ruxolitinib induction therapy (= baseline), at confinement to Ruxolitinib continuous therapy and after confinement at 6 months, 1 year, 2 years and 3 years
Overall Survival | 3 years
  Overall survival at 3 years after allogeneic SCT compared to Ruxolitinib continuous therapy in patients without a suit-able donor

CONTACTS AND LOCATIONS:
Overall Officials: Nicolaus Kröger, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (14):
- Germany (14):
  - Universitätsklinkum Aachen, Aachen
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinkum Halle, Halle
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Jena, Jena
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Johannes Wesling Klinikum Minden, Minden
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg, Nuremberg
  - Robert-Bosch-Krankenhaus Stuttgart, Stuttgart
  - Universitätsmedizin Tübingen, Tübingen
  - Universitätsklinkum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No